CLINICAL TRIAL: NCT04358289
Title: Generating Collective Solutions to Reduce Unnecessary Antibiotic Use in Vietnam
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 30HN
Record Dates: First submitted 2020-04-03; First posted 2020-04-24 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Antibiotic Use
Keywords: AMR; primary health care; Antimicrobial resistance
MeSH Terms: interventions — Residence Characteristics; Hospitals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1: Control group (No Intervention): For commune health center and community
- Arm 2: Basic antimicrobial stewardship education (Other): For commune health center and community
  Interventions: Other: Basic antimicrobial stewardship education
- Arm 3: 3. Basic AS education + community education (Other): For commune health center and community
  Interventions: Other: Basic antimicrobial stewardship education; Other: Community education
- Arm 4: Education + participatory action research (Other): For commune health center and community
  Interventions: Other: Basic antimicrobial stewardship education; Other: Participatory action research group in commune health center and community; Other: Community education
- Hospital intervention (Other): For hospital: The hospital interventions will use quality improvement using a participatory action research approach to improve antibiotic stewardship. These activities will be evaluated through a before and after knowledge, attitudes and practice (KAP) survey, to assess whether or not the engagement activities had a measurable impact on knowledge and behaviour. There are not sufficient hospitals in the area to conduct a cluster randomized evaluation, so we will conduct a before and after survey, patient record review, and overall antibiotic use data from the Pharmacy Department
  Interventions: Other: Antimicrobial stewardship program in hospitals

INTERVENTIONS:
Other: Basic antimicrobial stewardship education — Commune health center: Revision of guidelines for antibiotic prescribing for respiratory infections in primary care, Training primary healthcare doctors in the application of the new guidelines
  Arms: Arm 2: Basic antimicrobial stewardship education; Arm 3: 3. Basic AS education + community education; Arm 4: Education + participatory action research
Other: Participatory action research group in commune health center and community — * Establish a participatory action research group
  * Engagement with the group through participatory action research involving problem identification, planning change strategies, implementing strategies, and evaluation
  Arms: Arm 4: Education + participatory action research
Other: Antimicrobial stewardship program in hospitals — The intervention activities in hospitals will include: training a health-worker in each of the participating hospitals to act as a facilitator or "activator"; forming an antibiotic stewardship group; meeting regularly and following an action-research cycle that includes problem identification, planning change strategies, implementing strategies, and evaluating strategies
  Arms: Hospital intervention
Other: Community education — Development of educational materials for the community and farmers; Disseminated of messages through posters, leaflets and local media channels
  Arms: Arm 3: 3. Basic AS education + community education; Arm 4: Education + participatory action research

SUMMARY:
The study aims to develop community-based interventions targetting inappropriate antibiotic dispensing and use behaviours in rural Vietnam and has 3 research components.

Community and primary healthcare interventions: The investigators will conduct a four-armed cluster randomised controlled trial. The first arm will be a control arm with no interventions. The second intervention arm will have a basic antimicrobial stewardship intervention, involving working with the Ministry of Health, Medical Services Administration to revise guidelines for antibiotic prescribing for acute respiratory infections (ARI) in primary care, and then training primary healthcare doctors in their use. The third intervention arm will have basic antimicrobial stewardship guidelines and training for primary healthcare doctors, plus educational materials for the community, disseminated through posters, leaflets and local media channels. The fourth intervention arm will use a participatory action research approach to engage primary healthcare doctors and communities, in addition to the basic guidelines and training materials. The participatory action research approach will train local facilitators to lead community and health-worker groups through a cycle of problem identification, strategy development, implementation and review, focusing on inappropriate human and small-scale agricultural use of antibiotics.

Hospital interventions: The investigators will work with Provincial and District Hospitals serving these communities to implement quality improvement cycles for antibiotic stewardship, also using a participatory action research approach. This will also follow a cycle of a cycle of problem identification, strategy development, implementation and review.

DETAILED DESCRIPTION:
1. Main research questions:

   1.2.1 Community interventions: Can educational and participatory action research interventions delivered in the community reduce the inappropriate use of antibiotics? 1.2.2 Primary healthcare interventions: Can educational and participatory action research interventions delivered in primary healthcare reduce prescription of antibiotics for patients with acute respiratory infections, outside of the research context? 1.2.3 Hospital interventions: Can participatory action research interventions delivered in hospitals improve antibiotic stewardship and reduce prescription of antibiotics?
2. OBJECTIVES 2.1 Community interventions: to evaluate the impact of educational and participatory action research interventions in communities on the proportion of the population reporting antibiotic use in the last month 2.2 Primary healthcare interventions: to evaluate the impact of antibiotic stewardship training and participatory action research interventions on the proportion of patients with ARI prescribed an antibiotic in routine primary health care 2.3 Hospital interventions: to evaluate the impact of quality improvement using a participatory action research approach on antibiotic stewardship and the proportion of patients receiving antibiotic treatment 2.4 Qualitative evaluation: to understand community processes and engagement with behaviour change interventions
3. STUDY DESIGN 3.1 Design 3.1.1 and 3.1.2 Community and primary healthcare interventions: The community and primary healthcare interventions will be evaluated together through a four-armed cluster-randomised controlled trial design, consisting of 16 communes in each arm, with interventions delivered either at the commune health centre, the community, or both. The goal of the evaluation is to assess whether or not the community and primary healthcare interventions had a measurable impact on knowledge and behaviour. Each of the three intervention arms will be done in 16 communes, and the investigators will select a further 16 communes as controls, where there will be no intervention activities. At the beginning of the project, the investigators will randomly allocate 64 communes to receive one of the three interventions or no intervention.

3.1.3 Hospital interventions: The hospital interventions will use quality improvement using a participatory action research approach to improve antibiotic stewardship. These activities will be evaluated through a before and after knowledge, attitudes and practice (KAP) survey, to assess whether or not the engagement activities had a measurable impact on knowledge and behaviour. There are not sufficient hospitals in the area to conduct a cluster randomized evaluation, so the investigators will conduct a before and after survey, patient record review, and overall antibiotic use data from the Pharmacy Department.

3.1.4 Qualitative evaluation: The goal of the qualitative evaluation is to understand the group processes and community and health-worker engagement with the action groups, how the engagement activities affect behaviour, and in what contexts they work better or worse, in order to develop a theory of change. The investigators will conduct in-depth interviews and participant observation in selected communities, and at each of the participating hospitals, during each of the four phases of the meeting cycle, in order to understand decision-making processes, as well as influential social and power dynamics in the groups. Participant observation is a method used in research where the investigators engage with people and document the information: investigators document what people said, what they did, how they interacted within a given setting.

3.2 Study location The target population for both phases will be the general resident population of two to three districts in Nam Dinh Province, covering 64 rural communes. Investigators at the National Institute for Hygiene and Epidemiology (NIHE), have longstanding connections and experience of working with communities in this region and will take the lead in developing relationships with Provincial representatives.

3.3 Communities and study participants Engagement with communities will be run through Women's Union and Farmers' Union groups. The Women's Union is a national organisation promoting the health and wellbeing of women and families in Vietnam, and has widespread coverage and membership at community-level. Women's Union groups are run by paid representatives and meet regularly. The Farmers' Union is also a national organisation that promotes good farming practices. Farmers' Union groups are also run by paid representatives and meet regularly. During the strategy development phase of group activities, groups will be encouraged to invite local stakeholders to participate, including community healthcare workers, primary healthcare workers, animal healthcare workers, and pharmacists.

3.4 Commune health centres Commune health centres (CHCs) deliver most primary care services and national targeted health programmes to the population, especially in rural and mountainous areas including hygiene, vaccinations, antenatal care, safe delivery and health education. Screening examination, treatment and referrals for CHC attendees are also provided. Regarding coverage of commune health network in Vietnam, 99% of communes have a health centre, 70% have a doctor; and 79.3% provide traditional medicine services13.

ELIGIBILITY:
For communities:

Inclusion criteria:

* Commune officials consent to take part;
* Have a commune population larger than 3000 individuals;
* Have active Women's Union and Farmers' Union groups with a paid commune-level representative;
* Commune health centre has a doctor;
* Commune health centre has electronic database.

Exclusion criteria:

* Urban areas with a low proportion of farmers or low utilisation of CHCs for primary healthcare.

For study participants:

Inclusion criteria:

* Participant is willing and able to give informed consent for participation in the study;
* Community members normally resident in the study commune (living in the study commune and resident for at least three months);

Exclusion criteria:

* No one will be actively excluded from participating in this population-based study.

For Commune Health Centers:

Inclusion criteria:

* Serve a commune population larger than 3000 individuals;
* Have an average caseload of at least 10 consultations per facility per week for ARI verified by checking the database system of the provincial centre for disease control and prevention (CDC) where the implementation study is being conducted;
* Health centre doctor is normally employed at the centre and has been there for at least three months.

Exclusion criteria:

* Low antibiotic prescription rate for ARI of below 40%.

For Patient records:

Inclusion criteria:

* All patients' anonymised records.

Exclusion criteria:

* Don't have national health insurance/not recorded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3315 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Community: Proportion of the population reporting antibiotic use in the last month | After the last interview/survey, up to 18 months since study implementation
Community: Proportion of the population with a mild respiratory illness in the last month who didn't seek medical consultation and treatment (at a health facility or a pharmacy) | After the last interview/survey, up to 18 months since study implementation
Community: Proportion of farmers reporting antibiotic use for their animals in the last month | After the last interview/survey, up to 18 months since study implementation
Primary healthcare: Proportion of patients aged 1 to 65 years, consulting for ARI, who are prescribed antibiotics | After the last interview/survey, up to 18 months since study implementation
Primary healthcare: Proportion of the population reporting antibiotic use in the last month | After the last interview/survey, up to 18 months since study implementation
Hospital: Proportion of patients receiving antibiotic treatment in the three months preceding the survey | After the last interview/survey, up to 18 months since study implementation

SECONDARY OUTCOMES:
Community: Proportion of the population who have heard about antibiotic resistance | After the last interview/survey, up to 18 months since study implementation
Community: Proportion of the population who can correctly define antibiotic resistance (from a list of options) | After the last interview/survey, up to 18 months since study implementation
Community: Proportion of the population who can correctly identify at least two human health behaviours that can lead to antibiotic resistance (from a list of options) | After the last interview/survey, up to 18 months since study implementation
Community: Average number of days of illness in the last month | After the last interview/survey, up to 18 months since study implementation
Community: Average number of days unable to do usual activities due to illness (e.g. absent from school/work/farm work) in the last month | After the last interview/survey, up to 18 months since study implementation
Community: Proportion of farmers who can correctly identify at least two farming behaviours that can lead to antibiotic resistance (from a list of options) | After the last interview/survey, up to 18 months since study implementation
Primary healthcare: The proportion of patients that consulted with ARI in the preceding year | After the last interview/survey, up to 18 months since study implementation
Primary healthcare: Prescription rates for ARI patients in the preceding year | After the last interview/survey, up to 18 months since study implementation
Primary healthcare: Proportion of patients receiving an antibiotic with the denominator being | After the last interview/survey, up to 18 months since study implementation
Primary healthcare: Proportion of patients receiving an antibiotic prescription by diagnosis, age, season, recorded fever, sex | After the last interview/survey, up to 18 months since study implementation
Primary healthcare: The proportion of patients referred to a higher-level facility at the initial consultation by checking the e-database of health insurance (HI) reimbursement | After the last interview/survey, up to 18 months since study implementation
Hospital: Changes in knowledge and perceptions pf doctors in the month before the intervention starts, and the last month of intervention implementation | After the last interview/survey, up to 18 months since study implementation
  Based on a knowledge, attitude and practice survey.
Hospital: Proportion of patients receiving appropriate antibiotic treatment in the three months preceding the survey (Days of Therapy) | After the last interview/survey, up to 18 months since study implementation
Hospital: Number and proportion of patients whose antibiotic therapy was reviewed with feedback to the treating doctor by the stewardship team per month | After the last interview/survey, up to 18 months since study implementation
Hospital: Proportion of patients who had samples taken for culture before antibiotic initiation (where available) | After the last interview/survey, up to 18 months since study implementation
Hospital: Proportion of patients who received targeted antibiotic groups as empiric or culture adjusted therapy | After the last interview/survey, up to 18 months since study implementation
Hospital: Proportion of patients who had de-escalation after culture results were available | After the last interview/survey, up to 18 months since study implementation
Hospital: Proportion of patients who received appropriate antibiotic therapy after culture results were available | After the last interview/survey, up to 18 months since study implementation
Hospital: Count and proportion of resistant isolates for priority antibiotic-organism combinations (where available) | After the last interview/survey, up to 18 months since study implementation
Hospital: Cost of antibiotic treatment (Total monthly cost by department) | After the last interview/survey, up to 18 months since study implementation
Hospital: Cost of antibiotic treatment (Average cost per patient) | After the last interview/survey, up to 18 months since study implementation
Hospital: In-hospital mortality (Departmental wide) | After the last interview/survey, up to 18 months since study implementation
Hospital: In-hospital mortality (Patients receiving antibiotics) | After the last interview/survey, up to 18 months since study implementation
Hospital: Hospital length of stay | After the last interview/survey, up to 18 months since study implementation
The number of meetings that subject participates in Participatory Action Group 's meetings | After the last interview/survey, up to 18 months since study implementation

CONTACTS AND LOCATIONS:
Locations (1):
- Nam Dinh province, Nam Định, Vietnam